CLINICAL TRIAL: NCT04501549
Title: Plaque mOrphology iMpact on Side Branch Occlusion at oPtical Coherence Tomography Evaluation in Percutaneous Coronary Interventions: The POMPEI Study
Brief Title: Plaque mOrphology iMpact on Side Branch Occlusion at oPtical Coherence Tomography Evaluation in Percutaneous Coronary Interventions
Acronym: POMPEI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/2493
Record Dates: First submitted 2020-08-02; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Bifurcation; Percutaneous Coronary Intervention
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: percutaneous coronary intervention — PCI will be performed according to local practice.The bifurcation lesion will be imaged by OCT on at least two time-points for each patient. Plaque morphology will be characterized by OCT. Off-line quantitative coronary angiography (QCA) will be performed before and after PCI and the following QCA parameters will be computed: reference vessel diameter (RVD), lesion length and diameter stenosis (DS) of Main Vessel (MV) and side branch (SB). Blood samples will be taken prior to PCI and 8-12 hours later to determine peri-procedural myocardial injury and infarction following PCI by measuring serum Troponin.

SUMMARY:
Despite recent advances in interventional cardiology, bifurcation coronary artery stenoses (which account for 15-20% of all coronary lesions treated by PCI), remain a challenge for PCI operators with higher rates of failure, in-stent restenosis, stent thrombosis, and recurrent clinical events, when compared to simple non-bifurcation lesions.

POMPEI trial is a prospective observational study. We aim to investigate the impact of morphological plaque characteristics assessed by optical coherence tomography (OCT) on the risk of developing side branch occlusion (SBO) in bifurcation PCI.

A total of 27 patients undergoing bifurcation PCI will be recruited into the trial. PCI will be performed according to local practice.The bifurcation lesion will be imaged by OCT on at least two time-points for each patient. Plaque morphology will be characterized by OCT. Off-line quantitative coronary angiography (QCA) will be performed before and after PCI and the following QCA parameters will be computed: reference vessel diameter (RVD), lesion length and diameter stenosis (DS) of Main Vessel (MV) and side branch (SB). Blood samples will be taken prior to PCI and 8-12 hours later to determine peri-procedural myocardial injury and infarction following PCI by measuring serum Troponin. The OCT data analysis will be performed in collaboration with Dr Valeria Paradies who has been trained in interventional cardiology in Rotterdam (The Netherlands) with specific interest in intravascular imaging.

In conclusion, we will use OCT to detect specific morphological characteristics which are associated with acute SBO following main vessel stenting. The routine use of OCT during bifurcation PCI to detect those patients at risk of acute SBO following main vessel stenting will allow the PCI operator to implement measures for reducing the risk of SBO, thereby minimizing the risk of peri- and post-PCI angina, preventing peri-procedural myocardial injury and infarction, and improving clinical outcomes.

DETAILED DESCRIPTION:
We hypothesized that in bifurcation lesion treatment, morphology of the plaque located in the main vessel may impact on the risk of developing SBO.

The objectives of POMPEI study as follows:

Primary objective:

To identify correlation between lipid volume content of MV plaque and risk of SBO (TIMI flow<3)

Secondary objectives:

To identify the plaque morphology characteristics associated with SBO in patients undergoing bifurcation PCI. OCT parameters which will be assessed include: distribution of lipid volume and lipid arc in the MV and around SB ostium before and after stenting; prevalence of healed plaque rupture and erosion and its correlation with SBO; correlation between calcium distribution within the plaque and SBO; correlation between bifurcation angle and SBO; and correlation between angiographic images of haziness at SB ostium and OCT findings.

To determine the prevalence of significant SB ostium stenosis in patients undergoing bifurcation PCI.

To determine the incidences of SBO following bifurcation PCI.

To determine the incidence and extent of peri-procedural myocardial injury and infarction following bifurcation PCI.

To determine correlation between SB lesion extension from the ostium and SBO

ELIGIBILITY:
Inclusion Criteria:

* Age≥21 years of age
* Able to provide consent
* At least one de-novo bifurcation lesion involving a side-branch (SB) ≥ 2mm and SB ostial lesion ≥50% and <90% by visual assessment intended to be treated by PCI with provisional stenting strategy
* TIMI flow 3 in both MV and SB

Exclusion Criteria:

* Previous PCI of the target vessel
* Cardiac arrest or cardiogenic shock
* Left main or saphenous venous graft bifurcation
* Significant renal impairment patients (eGFR<30) who are not on dialysis
* Inability to advance the OCT catheter or to obtain good image quality

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient waiting lists will be screened for patients undergoing election PCI for known bifurcation lesions. Patients will also be recruited after the elective PCI procedure. Patients who have undergone elective PCI for a bifurcation lesion which fits the criteria below, and had OCT performed during the procedure for clinical reasons.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2021-04-14 (Estimated); Study Completion 2021-04-14 (Estimated)

PRIMARY OUTCOMES:
To undertake a proof-of-concept clinical study to investigate the impact of morphological plaque characteristics on the risk of developing SBO in bifurcation lesion treatment | 1year
  If we can show that different culprit plaques behave differently, then there is the potential to undertake a larger study to change the way we manage these plaques and therapies to prevent SBO.

CONTACTS AND LOCATIONS:
Overall Officials: Chin Chee Yang, MD, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore